CLINICAL TRIAL: NCT04133116
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3471851 in Japanese and Caucasian Healthy Subjects
Brief Title: A Study of LY3471851 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17414; J1P-MC-KFAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3471851 (Experimental): Participants received single doses of 450 microgram (μg), 900 μg or 1800 μg LY3471851 administered subcutaneously (SC).
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Placebo matching LY3471851 administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — Administered SC
  Other Names: NKTR-358
  Arms: LY3471851
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to explore the safety and tolerability of LY3471851 in healthy Japanese and Caucasian participants. The study will also estimate how much LY3471851 gets into the blood stream and how long it takes the body to remove it. The study is expected to last about 7 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females, as determined by medical history and physical examination
* Are first generation Japanese or are Caucasian
* Have a body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive, at the time of screening

Exclusion Criteria:

* Are currently enrolled in a clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have an abnormal blood pressure and/or pulse rate as determined by the investigator
* Regularly use known drugs of abuse and/or show positive findings on drug screening
* Are immunocompromised per investigator judgment

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Study Completion (up to week 7)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3471851 | Predose on Day 1 through Day 50
  PK: AUC of LY3471851
PK: Maximum Concentration (Cmax) of LY3471851 | Predose on Day 1 through Day 50
  PK: Cmax of LY3471851

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No